CLINICAL TRIAL: NCT01908101
Title: Phase II Trial of Metronomic Eribulin (Halaven) in Pretreated Metastatic Breast Cancer (MBC)
Brief Title: Eribulin Mesylate in Treating Patients With Previously Treated Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8093; NCI-2013-01326 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8093 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2013-07-19; First posted 2013-07-25 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-05

CONDITIONS: Recurrent Breast Carcinoma; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (eribulin mesylate) (Experimental): Patients receive eribulin mesylate IV over 2-5 minutes on days 1, 8, and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Eribulin Mesylate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Eribulin Mesylate — Given IV
  Other Names: B1939 Mesylate; E7389; ER-086526; Halaven; Halichondrin B Analog
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well eribulin mesylate works in treating patients with previously treated breast cancer that has spread to other places in the body. Drugs used in chemotherapy, such as eribulin mesylate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Progression free survival (PFS).

SECONDARY OBJECTIVES:

I. Frequency of alopecia with absence or decrease to < 50%.

II. Incidence of grade 3 and 4 neutropenia of < 30%.

III. Incidence of sensory neuropathy (all grades) to < 25%.

TERTIARY OBJECTIVES:

I. Assess the role of circulating endothelial cell precursors (CEPs) and apoptotic circulating endothelial cells (CECs), in predicting early response to treatment.

OUTLINE:

Patients receive eribulin mesylate intravenously (IV) over 2-5 minutes on days 1, 8, and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Prior exposure to taxane in the adjuvant, neoadjuvant or metastatic setting
* At least one prior regimen of chemotherapy in the setting of metastatic breast cancer; no upper limit on the number of prior endocrine regimens for metastatic breast cancer, however no more than 6 chemotherapeutic regimens may have been given in the metastatic setting
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patients must have baseline imaging within 30 days prior to the start of therapy and satisfy one of the following:

  * Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
  * At least one non lymph node lesion of >= 1.0 cm or lymph node >= 1.5 cm in short axis by computerized tomography (CT) scan (CT scan thickness no greater than 5 mm which is serially measurable according to RECIST 1.1 using either computerized tomography (CT) or magnetic resonance imaging (MRI)
  * Lesions that have had radiotherapy must show evidence of progressive disease (PD) based on RECIST 1.1 to be deemed a target lesion
  * Non-measurable disease by RECIST 1.1 criteria (includes bone only disease and lesions < 10 mm or lymph nodes < 15 mm in short axis) with rising serum CA15-3 or CA 27.29 or CEA documented by two consecutive measurements taken at least 14 days apart with the most recent measurement being within 42 days prior to registration. The second CA 15-3 or CA 27.29 value must have at least a 20% increase over the first and for CA 15-3 or CA27.29 be greater than or equal to 40 units/mL or for CEA be greater than or equal to 4 ng/mL
* Absolute neutrophil count >= 1,500/mm^3
* Hemoglobin >= 10 g/dL
* Platelets >= 100,000/mm^3
* Creatinine =< 1.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN
* Alkaline phosphatase =< 3.0 x ULN; up to 5 x ULN is acceptable if due to bone metastases in the absence of liver metastases
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x institutional upper limit of normal, unless due to liver metastases (=< 5 x ULN)
* Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation
* Life expectancy of > 12 weeks

Exclusion Criteria:

* Prior treatment with eribulin
* Plan to administer any other systemic antitumor including endocrine therapy except for following standard of care treatment:

  * Trastuzumab at standard dosing human epidermal growth factor receptor 2 (HER2) positive tumors
  * Denosumab or bisphosphonates to treat metastatic bone disease
* Plan to administer concurrent radiation therapy now or for progressive symptoms during treatment
* Patients with known central nervous system (CNS) metastases must have stable disease off steroids after treatment with surgery or radiation therapy
* Second primary malignancy that is clinically detectable or clinically significant at the time of consideration for study enrollment
* Patients with mild (Child-Pugh A) or moderate (Child-Pugh B) hepatic and/or moderate (creatinine clearance [CrCl] 30-50 mL/min) renal impairment
* Radiotherapy within 14 days of study treatment
* Major surgery within 21 days of study treatment; minor surgery within 2 weeks of study treatment; placement of vascular access device and biopsies allowed and is not considered major or minor surgery
* Treatment with any systemic chemotherapy or investigational agents within 3 weeks of the start of study treatment; endocrine treatment must be stopped prior to initiating study treatment; subjects must have recovered from toxicities of prior therapy
* Patients with peripheral neuropathy > grade 2 regardless of etiology
* Significant cardiovascular impairment: congestive heart failure > class II according to the New York Heart Association (NYHA), unstable angina or myocardial infarction within 6 months of enrollment, or serious cardiac arrhythmia (> grade 2)
* Concomitant severe or uncontrolled medical disease
* Significant psychiatric or neurologic disorder which would compromise participation in the study
* Pregnant or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2019-05-04 (Actual); Study Completion 2019-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Linden, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (12):
- United States (12):
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Bend Memorial Clinic, Bend, Oregon
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 86 patients signed the study informed consent, but only 68 patients started the Eribulin treatment. Out of those 68 patients only 59 of them were evaluable.
Period: Overall Study
Arm/Group | Treatment (Eribulin Mesylate)
Started | 68
Completed | 59
Not Completed | 9
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Incorrect Diagnosis | 2
Not completed — Incorrect Starting Dose | 1
Not completed — Did not complete the first cycle | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 52 [18 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: PFS
Description: Kaplan-Meier survival curves will be used to describe PFS, overall and stratified by number of prior metastatic treatment regimens. A 95% confidence interval for the median PFS will be calculated using the method of Brookmeyer and Crowley.
Time Frame: From study enrollment until the earliest date of disease progression or death, assessed up to 1 year
Population: Patients with metastatic breast cancer (MBC) whose disease has progressed following at least one prior regimen of chemotherapy in the setting of metastatic breast cancer
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 59
months | 3.5 [2.6 to 4.6]
Statistical Analysis 1: Comparison: Treatment (Eribulin Mesylate); Progression free survival (PFS). We hypothesize that metronomic dosing of eribulin will result in a PFS of 4-6 months; Test type: Other — comparison analysis; comparison analysis; no P value; Median Difference (Final Values) = 3.5, 95% CI 2-sided [2.6 to 4.6] — The estimated value is 3.5 months, not years

ADVERSE EVENTS:
Time Frame: Adverse events will be collected after the patient has taken the first dose of study drug. After discontinuation from treatment, patients must be followed for all existing AEs for 30 calendar days after the last dose of study drug or until another anti-cancer therapy is initiated.
Arm/Group | Treatment (Eribulin Mesylate)
All-Cause Mortality (participants affected / at risk) | 44/59
Serious Adverse Events (participants affected / at risk) | 2/59
Other Adverse Events (participants affected / at risk) | 23/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Eribulin Mesylate) (N=59)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Eribulin Mesylate) (N=59)
Fatigue (General disorders) | 3 (3)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Nervous system disorders) | 13 (13)
Peripheral neuropathy (Nervous system disorders) | 3 (3)
White blood cell decreased (Blood and lymphatic system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT01908101/Prot_SAP_000.pdf